CLINICAL TRIAL: NCT03066999
Title: Assessment of the Effectiveness and Ease of Use of DirectVision- a Direct Visualization System for Urinary Catheterization: Results of a Single Center Prospective Study
Brief Title: DirectVision for Urinary Catheterization
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: There was no enough subject
Sponsor: The Pur Clinic (Other)
Collaborators: PercuVision (Unknown)
Responsible Party: Principal Investigator, Sijo J. Parekattil, M.D., Director of PUR clinic, Investigator, The Pur Clinic
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: 16.129.10
Record Dates: First submitted 2017-02-08; First posted 2017-03-01 (Actual); Results first posted 2019-07-30 (Actual); Last update posted 2019-07-30 (Actual); Status verified 2019-07

CONDITIONS: Urethral Diseases
MeSH Terms: conditions — Urethral Diseases | interventions — Cystoscopy

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (2):
- Cystoscopy (Active Comparator): will have catheter placement using the cystoscopy method
  Interventions: Procedure: Cystoscopy
- DirectVision (Active Comparator): will have catheter placement using DirectVision.
  Interventions: Device: DirectVision

INTERVENTIONS:
Procedure: Cystoscopy — Patients will assign to either Group Cystoscopy (catheter placement via cystoscopy)
  Arms: Cystoscopy
Device: DirectVision — Patients will assign to either Group DirectVision (catheter placement via DirectVision)
  Arms: DirectVision

SUMMARY:
The Center for Disease Control and Prevention (CDC) reports that one in four patients hospitalized in the United States is catheterized to void the bladder or monitor urinary output. In the male population, Dr. Singh, an urologist estimates that about 20% of catheterizations are difficult. Driving a catheter blindly, guessing whether to push the catheter forward or manipulate it to get around a point of resistance leads to the risk of injury which increases the more the catheter is manipulated. Additional adverse events include: urosepsis, UTI and bladder perforation. The standard of care treatment for patients with difficult urinary catheterization (DUC) is to proceed with a cystoscopic catheter placement or suprapubic tube placement.

PercuVision has the only Foley catheter with a micro-endoscope for visualization and navigation of the urethra for nurses and other qualified health care professionals. Moreover, it allows urologists to place a guidewire under direct vision rather than calling for a flexible cystoscope which is considered a minor procedure.

In this study, the investigators plan on assessing the effectiveness and ease of use of the PercuVision DirectVision® System device.

DETAILED DESCRIPTION:
Routine placement of transurethral catheters can be challenging in some situations, such as urethral strictures, severe phimosis and false passages. Intravaginal retraction of the urethral meatus can complicate Foley placement in postmenopausal females. In men, blind urethral procedures with mechanical or metal sounds without visual guidance or guidewire assistance are now discouraged due to the increased risk of urethral trauma and false passages.

DirectVision is a new visually-guided catheterization device (VGCD) that uses a camera visual guide / microendoscope within a triple lumen flexible urinary catheter with an angled tip, essentially combining the functionality of a urinary catheter with a cystoscope. DirectVision uses fiber-optic bundle of 6,000 integrated fibers to provide illumination and transmit real-time video.

Procedures done via flexible cystoscopy or DirectVision are covered by insurance (including Medicaid/Medicare).

In this prospective study, the investigators plan on assessing the effectiveness and ease of use of DirectVision - A direct visualization system for urinary catheterization.

ELIGIBILITY:
Inclusion Criteria:

* Any patient over 18 years with a standard indication for difficult urinary catheterization

Exclusion Criteria:

* Any patient younger than 18 years of age, pregnant patients

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 5 (Actual)
Dates: Start 2017-03-07 (Actual); Primary Completion 2017-10-01 (Actual); Study Completion 2017-10-01 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- South Lake Hospital, Clermont, Florida, United States

IPD SHARING:
Plan to Share IPD: No
We will keep the IPD within the research group

REFERENCES:
- [Background] Ghaffary C, Yohannes A, Villanueva C, Leslie SW. A practical approach to difficult urinary catheterizations. Curr Urol Rep. 2013 Dec;14(6):565-79. doi: 10.1007/s11934-013-0364-3. PMID 23959835
- See also: Feasibility study of a visually guided male urinary catheterization device by Banks et al.Journal of Urology. 2009; 181(4): p454. — https://www.researchgate.net/publication/246174153_FEASIBILITY_STUDY_OF_A_VISUALLY_GUIDED_MALE_URINARY_CATHETERIZATION_DEVICE

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: No enrolled patients were excluded from the study before assignment to groups
Groups:
- Cystoscopy: Patient will have catheter placement using the cystoscopy method
- DirectVision: Patient will have catheter placement using DirectVision.
Period: Overall Study
Arm/Group | Cystoscopy | DirectVision
Started | 2 | 3
Completed | 2 | 1
Not Completed | 0 | 2
Not completed — abnormal urethraBladder neck contracture | 0 | 2

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Cystoscopy | DirectVision | Total
Number analyzed (Participants) | 2 | 3 | 5
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 0 | 0 | 0
  >=65 years | 2 | 3 | 5
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 0 | 0
  Male | 2 | 3 | 5
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
History of urological procedures [Count of Participants; unit: Participants] | 2 | 2 | 4

OUTCOME MEASURES:

1. Primary Outcome: Set up Time/Total Procedure Time to Place Catheter Via DirectVision/Cystoscope
Description: Duration to set up and complete the procedure either by DirectVision or Cystoscope was observed and calculated by minutes.
Time Frame: prep and duration of procedure, up to 1 hour
Measure: Mean (Full Range); unit: minutes
Groups:
- Cystoscopy: will have catheter placement using the cystoscope
Arm/Group | Cystoscopy | DirectVision
Number analyzed (Participants) | 2 | 3
minutes
  Set up time- in minutes | 15 [15 to 15] | 26.67 [20 to 30]
  procedure time | 5 [5 to 5] | 23.33 [10 to 30]

2. Primary Outcome: Effectiveness of DirectVision-adverse Events
Description: assessment will be done by reviewing the number of Participants who had adverse events that are related to the procedures.
Time Frame: 7 months
Measure: Count of Participants; unit: Participants
Arm/Group | Cystoscopy | DirectVision
Number analyzed (Participants) | 2 | 3
Participants | 0 | 0

3. Primary Outcome: Ancillary Tools Used
Description: Ancillary tools used wire, SPT, etc
Time Frame: duration of procedure
Measure: Number; unit: tools
Arm/Group | Cystoscopy | DirectVision
Number analyzed (Participants) | 2 | 3
tools | 2 | 2

4. Primary Outcome: Procedure Findings
Description: Procedure findings
  * 1- Obliterated urethra
  * 2-High bladder neck
  * 3-Normal urethra
  * 4-Urethral stricture
  * 5-Bladder neck contracture
Time Frame: duration of procedure
Measure: Number; unit: participants
Arm/Group | Cystoscopy | DirectVision
Number analyzed (Participants) | 2 | 3
participants
  Obliterated urethra | 0 | 1
  High bladder neck | 1 | 0
  Normal urethral profile | 0 | 1
  Urethral stricture | 1 | 0
  Bladder neck contracture | 0 | 1

5. Primary Outcome: Degree of Difficulty
Description: Degree of difficulty defined as easy versus difficult
Time Frame: duration of procedure
Measure: Count of Participants; unit: Participants
Arm/Group | Cystoscopy | DirectVision
Number analyzed (Participants) | 2 | 3
Participants
  Easy | 2 | 1
  Difficult | 0 | 2

6. Primary Outcome: Presence of Pain and Hematuria
Description: To compare DirectVision to the cystoscope we compared if patients experienced pain or hematuria
Time Frame: duration of procedure
Measure: Number; unit: participants
Arm/Group | Cystoscopy | DirectVision
Number analyzed (Participants) | 2 | 3
participants
  Presence of hematuria | 1 | 1
  Presence of pain | 0 | 0

7. Secondary Outcome: Cost to Use Cystoscope Versus DirectVision
Description: The investigators will look at the cost using the DirectVision versus the cystoscope with costs of ancillary tools used during the procedures.
Time Frame: 7 months
Measure: Mean (Full Range); unit: Cost in dollars per patient
Arm/Group | Cystoscopy | DirectVision
Number analyzed (Participants) | 2 | 3
Cost in dollars per patient | 174 [174 to 174] | 187 [164 to 198]

ADVERSE EVENTS:
Time Frame: From procedure through discharge from hospital
Description: No adverse event noted
Arm/Group | Cystoscopy | DirectVision
All-Cause Mortality (participants affected / at risk) | 0/2 | 0/3
Serious Adverse Events (participants affected / at risk) | 0/2 | 0/3
Other Adverse Events (participants affected / at risk) | 0/2 | 0/3

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2017-02-28): https://cdn.clinicaltrials.gov/large-docs/99/NCT03066999/Prot_SAP_000.pdf
  • Informed Consent Form (2017-07-26): https://cdn.clinicaltrials.gov/large-docs/99/NCT03066999/ICF_001.pdf